CLINICAL TRIAL: NCT02310295
Title: Bevacizumabe e Acetato de Triancinolona Intra-vítreo Associados à Laserterapia em Pacientes Com Edema Macular diabético (IBeTA)
Brief Title: Prospective, Randomized Clinical Trial Comparing Macular Photocoagulation With or Without Intravitreal Bevacizumab or Triamcinolone for the Treatment of Diabetic Macular Edema
Acronym: IBeTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Messias, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12029-2008
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic retinopathy; Macular edema; Anti-VEGF; Triamcinolone
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Lasers; Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IVB-Laser (Active Comparator): Intravitreal Bevacizumab combined with focal laser therapy
  Interventions: Device: Laser; Drug: Bevacizumab
- IVTA-Laser (Active Comparator): Intravitreal Triamcinolone combined with focal laser therapy
  Interventions: Device: Laser; Drug: Triamcinolone Acetonide
- Laser (Active Comparator): focal laser therapy
  Interventions: Device: Laser

INTERVENTIONS:
Device: Laser — focal macular laser therapy
Drug: Bevacizumab — Intravitreal injection of Bevacizumab
  Arms: IVB-Laser
Drug: Triamcinolone Acetonide — Intravitreal injection of Triamcinolone Acetonide
  Arms: IVTA-Laser

SUMMARY:
Purpose: To compare the effects of macular photocoagulation with or without intravitreal bevacizumab (IVB) or triamcinolone (IVTA) for the treatment of diabetic macular edema (DME). Casuistic and Methods: 58 eyes of 44 patients with diffuse DME were randomized to receive either IVB + focal/grid laser (IVB-Laser, n=19), IVTA + focal/grid laser (IVTA-Laser, n=16) or focal/grid laser alone (Laser, n=23). Ophthalmic evaluation, including best-corrected visual acuity (BCVA), intraocular pressure (IOP) and central macular thickness (CMT) were performed at baseline and monthly for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. clinically significant diabetic macular edema (DME) with diffuse leakage involving the center of the fovea, with DME greater than 275 microns in OCT examination
2. BCVA between 0.3 LogMAR (logarithm of smaller angle of visual resolution) (20/40) and 1.6 LogMAR (20/800)
3. signed of inform Consent.

Exclusion Criteria:

1. HbA1c levels greater than 10%
2. thromboembolic event history (including myocardial infarction and stroke)
3. vitreo-macular traction on OCT
4. coagulation disorders
5. macular ischemia on fluorescein angiography examination
6. proliferative diabetic retinopathy that required treatment
7. eye surgery
8. history of ocular hypertension or glaucoma
9. any ocular pathology which in the opinion of the investigator, could macular edema or change the visual acuity during the study period (for example, retinal vascular occlusion, uveitis or other inflammatory eye disease, neovascular glaucoma)
10. systemic corticosteroid therapy
11. any conditions that could affect the documentation
12. any previous treatment for diabetic macular edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Central subfield macular thickness | 12 months
  retinal thickness measured with optical coherence tomography
Visual acuity | 12 months
  Best corrected visual acuity